CLINICAL TRIAL: NCT02209779
Title: A Randomised, Parallel, Double-blind, Placebo-controlled Study to Investigate Efficacy and Safety of Different Doses (5, 10, 20 and 30 mg) of BIRB 796 BS Administered Twice a Day Orally Over 4 Weeks in Patients With Active Rheumatoid Arthritis Who Have Failed at Least One DMARD
Brief Title: Efficacy and Safety of Different Doses of BIRB 796 BS in Patients With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1175.11
Record Dates: First submitted 2014-08-05; First posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid

ARMS (5):
- BIBR 796 BS, low dose (Experimental): twice daily doses of 5 mg for 4 weeks
  Interventions: Drug: BIBR 796 BS; Drug: Placebo
- BIBR 796 BS, medium dose 1 (Experimental): twice daily doses of 10 mg for 4 weeks
  Interventions: Drug: BIBR 796 BS; Drug: Placebo
- BIBR 796 BS, medium dose 2 (Experimental): twice daily doses of 20 mg for 4 weeks
  Interventions: Drug: BIBR 796 BS; Drug: Placebo
- BIBR 796 BS, high dose (Experimental): twice daily doses of 30 mg for 4 weeks
  Interventions: Drug: BIBR 796 BS
- Placebo (Active Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIBR 796 BS
  Arms: BIBR 796 BS, high dose; BIBR 796 BS, low dose; BIBR 796 BS, medium dose 1; BIBR 796 BS, medium dose 2
Drug: Placebo
  Arms: BIBR 796 BS, low dose; BIBR 796 BS, medium dose 1; BIBR 796 BS, medium dose 2; Placebo

SUMMARY:
The objective was to determine the effects of BIRB 796 BS on CRP and clinical parameters in Rheumatoid Arthritis as measures of efficacy, and on population pharmacokinetics and safety parameters

ELIGIBILITY:
Inclusion Criteria:

* Male or female from 18 to 75 years of age
* Diagnosis of Rheumatoid Arthritis (RA) established according to ACR criteria and date of diagnosis >1 year to ≤ 15 years. The exclusion of patients with a disease duration > 15 years was deleted in Amendment 2, effective January 22, 2002
* Patient belonging to functional class I, II, or III
* Failure of at least one Disease Modifying Antirheumatic Drug (DMARD) due to inefficacy
* Active disease, documented at visit 3, defined by ≥10 swollen joints in a 66 joint count and ≥ 12 tender joints in a 68 joint count
* CRP ≥ 2.0 mg/dl at visit 1 or visit 2
* Written informed consent in accordance with Good Clinical Practice and local legislation given prior to any study procedures, including washout of prohibited medications

Exclusion Criteria:

* Pregnancy (to be excluded by serum and urine β Human Chorion-Gonadotropin-test in women of childbearing potential) or breast feeding
* Female of childbearing potential (not 6 months post-menopausal or surgically sterilized) not using an approved form of birth control (hormonal contraceptives, oral or injectable/implantable, intra-uterine device (IUD))
* Inflammatory rheumatic disease other than RA
* Active vasculitis or any history of vasculitis (characterised by e.g. nail bed hemorrhages or infarcts, vasculitic purpura, ulcers or gangrenes, multisensory neuropathy, vasculitic retinopathy or scleritis of eyes). Isolated rheumatoid nodules of the skin are not a criterion for exclusion
* Treatment failure to a TNF-blocking agent. Treatment failure is defined as not achieving at least an ACR 20 response (e.g. in a clinical trial) or - in clinical practice - having the TNF-blocking agent discontinued due to ineffectiveness
* DMARD treatment within 4 weeks before visit 3
* Last dose given within the specified time period before visit 3 for one of the following compounds or drugs:

  * Infliximab (Remicade®): 3 months
  * D2E7 (a human TNF-α antibody): 3 months
  * Leflunomide (Arava®): 1 year, with exception of patients having undergone elimination therapy (colestyramin 8 grams t.i.d. po for eleven consecutive days), this exclusion criterion was deleted in Amendment 1, effective September 3, 2001
  * Drug classified as proton pump inhibitor: 7 days
  * Drug classified as H2-receptor-blocker or antacid: 2 days
  * Investigational agent: 5-fold of the respective plasma half life or 4 weeks, whichever is longer
* Treatment with systemic corticosteroids in a dose higher than 10 mg/day prednisone equivalent within 4 weeks prior to visit 3
* Change in treatment with nonsteroidal antiinflammatory drugs (NSAIDs) or systemic corticosteroids within 4 weeks prior to visit 3
* Synovectomy, joint surgery, radio-/chemo synoviorthesis or steroid injections (intraarticular, intravenous or intramuscular) within 4 weeks before visit 3
* Active infection or serious infectious diseases resulting in hospitalisation or requiring systemic anti-infective therapy within 4 weeks before visit 3
* Serologic evidence of active hepatitis B and/or C
* Known HIV-infection
* History of prior tuberculosis infection or suspicion of active infection at screening based on chest x-ray done within 6 month before visit 1
* History of cardiovascular, renal, neurologic, psychiatric, liver, gastrointestinal, immunologic or endocrine dysfunction if they are clinically significant. A clinically significant disease is defined as one which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study
* Recent history of heart failure, defined according to New York Heart Association criteria as being stage III or IV (i.e. three years or less) or myocardial infarction (i.e. one year or less) or patients with any cardiac arrhythmia requiring drug therapy. This exclusion criterion was slightly modified in Amendment 2, effective January 22, 2002.
* ECG results outside of the reference range of clinical relevance including, but not limited to QTcB > 480 msec, PR interval > 240 msec, QRS interval > 110 msec
* History of malignant disease in the last 5 years or suspicion of active malignant disease except successfully treated squamous or basal cell carcinoma of the skin
* Clinically significant abnormal baseline hematology, blood chemistry or urinalysis if the abnormality defines a disease listed as an exclusion criterion
* Any of the following specific laboratory abnormalities:

  * Alanine aminotransferase, aspartate aminotransferase, or total bilirubin greater than upper limit of normal (ULN) at visit 1 or measured within the last six months before visit 3. This exclusion criterion was modified in Amendment 1, effective September 3, 2001, allowing for a retest at Visit 2.
  * Gamma-Glutamyltransferase, alkaline phosphatase or Lactate Dehydrogenase greater than 1.5 x ULN at visit 1
  * creatinine or white blood cell count greater than 1.5 x ULN at visit 1
* History of drug or alcohol abuse within the past two years or active drug or alcohol abuse, present alcohol intake more than three drinks per day
* Inability to comply with the protocol
* Participation in another clinical trial within 30 days before visit 3
* Previous enrolment in this trial
* Hypersensitivity to trial drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2001-05; Primary Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
Absolute difference to baseline in concentrations of C-reactive Protein (CRP) | before and after 4 weeks of treatment

SECONDARY OUTCOMES:
Absolute difference to baseline in tender joint count (TJC, 68 joint count) | before and after 4 weeks of treatment
Absolute difference to baseline in swollen joint count (SJC, 66 joint count) | before and after 4 weeks of treatment
Patients assessment of pain on a visual analogue scale (VAS) | up to 57 days
Patients global assessment of disease activity (PADA) on a VAS | up to 57 days
Physicians global assessment of disease activity on a VAS | up to 57 days
Assessment of physical function by a standardised health assessment questionnaire (HAQ) | up to 57 days
Absolute difference to baseline in Erythrocyte sedimentation rate (ESR) | up to 57 days
Absolute difference to baseline in Cytokines Tumor Necrosis Factor (TNF)-α, soluble TNF-Receptor (sTNF-R), Interleukin (IL)-1ra, IL-6 | Day 1, 8 and 29
Absolute difference to baseline in Matrix metalloprotease-3 (MMP-3) | Day 1, 8 and 29
Absolute difference to baseline in Vascular endothelial growth factor (VEGF) | Day 1, 8 and 29
Number of responders to American College of Rheumatology (ACR) preliminary response criteria for 20% improvement (ACR 20), ACR 50, ACR 70 | after 4 weeks of treatment
Number of responders to European League against Rheumatism (EULAR) response criteria | after 4 weeks of treatment
Number of drop-outs due to lack of efficacy, according to final assessment of investigator | after 4 weeks of treatment
Assessment of maximum concentration (Cmax) | Day 15, 22, 29
Assessment of area under the curve (AUC) at steady state | Day 15, 22, 29
Number of patients with Adverse events | up to day 73